CLINICAL TRIAL: NCT03646500
Title: Prospective Randomized Controlled Trial Comparing Conscious Sedation to Retrobulbar Block Anesthetics During Trans-scleral Diode Laser
Brief Title: Comparing Conscious Sedation to Retrobulbar Block Anesthetics During Trans-scleral Diode Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Delan Jinapriya, Assistant Professor (Dept. of Ophthalmology); Eye Physician and Surgeon; Glaucoma Subspecialist, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18096
Record Dates: First submitted 2015-09-21; First posted 2018-08-24 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled non-inferiority trial, with retrobulbar block being the gold standard. Patients will be randomized to receive conscious sedation or retrobulbar injection prior to trans-scleral diode laser (TSD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retrobulbar block (Experimental): Retrobulbar block administered prior to Transcleral Diode Procedure
  Interventions: Procedure: Retrobulbar Block
- Remifentanil (Active Comparator): Conscious IV sedation administered prior to Transcleral Diode Procedure.
  Interventions: Procedure: Remifentanil

INTERVENTIONS:
Procedure: Retrobulbar Block — Anesthetic nerve block administered in the retrobulbar space prior to transcleral diode procedure
  Arms: Retrobulbar block
Procedure: Remifentanil — Remifentanil administered as intravenous infusion prior to transcleral diode procedure
  Other Names: remifentanil hydrochloride
  Arms: Remifentanil

SUMMARY:
This is a non-inferiority trial with a prospective randomized controlled design assessing patient satisfaction and complications associated with both retrobulbar block anesthetics (current gold standard) and conscious IV sedation alone (alternative choice of anesthesia) for trans-scleral diode laser (TSD). Patient satisfaction and complications will be measured using standardized patient surveys.

DETAILED DESCRIPTION:
This is a non-inferiority trial with a prospective randomized controlled design assessing patient satisfaction and complications associated with both retrobulbar block anesthetics (current gold standard) and conscious IV sedation alone (alternative choice of anesthesia) for trans-scleral diode laser (TSD). Patient satisfaction and complications will be measured using standardized patient surveys.

Methodology:

1. Patients undergoing TSD would be recruited from one glaucoma subspecialist's practice.
2. Patient consents to TSD at the eye clinic.
3. Clinical trial is mentioned to the patient and if there is interest a consent form is given to the patient to look over and develop questions the patient may want to ask.
4. Pre-anesthesia consult will be conducted to determine eligibility for both conscious sedation and retrobulbar block.
5. Patient is contacted by phone by the study coordinator to discuss whether the patient is still eligible to be a part of the clinical trial and whether the patient is still interested and if yes, what questions the patient might have. If the patient wishes to meet in person this will be arranged and consent can be obtained at that time, but if the patients are from a far distance then the signing of the consent will happen on the day of the procedure (although the discussion would already have taken place over the phone).
6. Patients will be randomized to either conscious sedation group, or retrobulbar injection group (control) via an online program.
7. On the day of the surgery, patients will receive a pre-anesthesia questionnaire (questions include basic identifying, health and surgery information).
8. Patients will receive a post-surgery questionnaire one hour after the surgery, in the recovery room.
9. Patients will receive a phone call for a post-recovery questionnaire 24 hours later.
10. Patients will receive a recovery and complications questionnaire one week later at the clinic (during check-up).

ELIGIBILITY:
Inclusion Criteria:

* ability to consent
* eligibility for both a conscious sedation and a retrobulbar block (decided through pre-anesthesia consult, which is a standard consult obtained for this procedure)

Exclusion Criteria:

* pregnancy
* inability to consent
* under 18 years of age
* not eligible for conscious sedation and/or retrobulbar block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Leiden Perioperative Care Patient Satisfaction Questionnaire | 1-week
  Self reported questionnaire measures patient satisfaction with perioperative care in the following dimensions: Information, Discomfort and Needs, Fear and Concern, Staff-Patient relationship, Service. Information, Staff-Patient Relationship scored as on a 5 point scale: Completely Satisfied, Dissatisfied, Not satisfied, nor dissatisfied, Satisfied, Completely Satisfied. Discomfort and needs and Fear and Concern are scored on a 5 point scale: Not at all, A little bit, Moderately, Quite a bit, Extremely).

SECONDARY OUTCOMES:
Core Measures of Outcomes of Anesthesia | 1-week
  Complication Rates

CONTACTS AND LOCATIONS:
Overall Officials: Delan Jinapriya, MD, Principal Investigator — Queen's University - School of Medicine
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided